CLINICAL TRIAL: NCT01878123
Title: A Randomized, Single-Dose, Placebo-Controlled, Study of the Safety, Tolerability, and Pharmacokinetics of AMP-110 in Subjects With Rheumatoid Arthritis
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of AMP-110 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMP-110-01
Record Dates: First submitted 2013-05-22; First posted 2013-06-14 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; Rheumatoid Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases; Antirheumatic agents
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMP-110 (Experimental): Escalating doses of AMP-110
  Interventions: Biological: AMP-110
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AMP-110 — Dose levels 1 through 7: Single intravenous infusion on Day 0
  Arms: AMP-110
Other: Placebo — Dose levels 4 through 7: Single intravenous infusion on Day 0
  Arms: Placebo

SUMMARY:
This is a Phase 1, single-dose, placebo-controlled, dose-escalation,multi-center, first time in human study of AMP-110 in adult subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide written informed consent
* Body mass index 18.5 to 35.0 kg/m2
* Diagnosis of Rheumatoid Arthritis according to 1987 revised American College of Rheumatology (ACR) criteria
* Global Functional Class I, II, or III according to ACR 1991 revised criteria
* Stable use of >/= 1 Disease Modifying Anti-rheumatic Drugs (DMARD) for >/= 4 weeks prior to Day 0, including:

  1. Methotrexate (MTX) 7.5 - 25 mg/week
  2. Hydroxychloroquine (HCQ) </= 400 mg/day
  3. Sulfasalazine (SSZ) 1,000 - 3,000 mg/day
  4. Leflunomide 5 - 20 mg/day
  5. Azathioprine 150 mg/day or 2 mg/kg/day
  6. Combinations of MTX, HCQ, and/or SSZ allowed

Exclusion Criteria:

* Prior to Day 0, use of

  1. Abatacept
  2. Rituximab within 6 months
  3. Infliximab, Adalimumab, Certolizumab, Tocilizumab, Cyclosporine, or Mycophenolate mofetil within 2 months
  4. Etanercept or Anakinra within 28 days
  5. Immunoglobulin or blood products within 28 days
* Evidence of any active or recent infection including ongoing, chronic infectious disease such as chronic renal infection or chronic chest infection with bronchiectasis or sinusitis
* History of systemic autoimmune disease other than Rheumatoid Arthritis
* History of allergic reactions to other protein therapeutics such as monoclonal antibodies or fusion proteins
* History of anaphylaxis or allergic diathesis
* Clinically significant cardiac disease, including: unstable angina; myocardial infarction within 6 months; congestive heart failure; arrhythmia requiring active therapy, with the exception of clinically insignificant extrasystoles, or minor conduction abnormalities; and history of clinically significant abnormality on electrocardiogram
* Evidence of active or latent tuberculosis
* Vaccination wtih live attenuated viruses within the 2 weeks prior to Day 0
* Evidence of infection with hepatitis B virus, hepatitis C virus, human immunodeficiency virus 1 or 2, or active infection with hepatitis A
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of a single dose of AMP-110 versus placebo | From start of study drug administration through Day 56
  Evaluate number of subjects with dose-limiting toxicities (through Day 14), evaluate number of subjects wtih adverse events (through Day 56), and number of subjects wtih changes from baseline in laboratory values, vital signs, physical exam and electrocardiogram (through Day 56)
Determine Maximum Tolerated Dose and/or recommended dose level(s) for future clinical trials | From start of study drug administration through Day 56
  Based on the occurrence of dose-limiting toxicities (through Day 14)

SECONDARY OUTCOMES:
Evaluate pharmacokinetic profile of a single dose of AMP-110 | From Day 0 pre-dose through Day 28
  Pharmacokinetics evaluated by area under the serum concentration versus time curve (AUC), peak serum concentration (Cmax), and clearance (Cl) of AMP-110

OTHER OUTCOMES:
Assess pharmacokinetic and pharmacodynamic relationships | From Day 0 pre-dose through Day 56
  Determine if pharmacodynamics effects of AMP-110 on certain cytokine levels and T cell subsets are dependent on serum drug concentrations
Evaluate exploratory biomarkers | From start of study drug administration through Day 56
  Blood samples will be analyzed throughout the study to characterize the physiological effects of AMP-110 treatment and to determine markers that correlate with response to treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas